CLINICAL TRIAL: NCT00198536
Title: Efficacy and Safety of Ecabet Ophthalmic Solution (2.83% and 3.70%) for Treatment of Dry Eye Syndrome
Brief Title: Efficacy and Safety Study for Ecabet Ophthalmic Solution for Treating Dry Eye Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-ECBT-CS01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ecabet 2.83% (Experimental): Ecabet ophthalmic solution One drop in study eye 4 times daily for 90 days.
  Interventions: Drug: Ecabet 2.83%
- Ecabet 3.70% (Experimental): Ecabet ophthalmic solution One drop in study eye 4 times daily for 90 days.
  Interventions: Drug: Ecabet 3.70%
- Vehicle (Placebo Comparator): One drop of vehicle in study eye 4 times daily for 90 days.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ecabet 2.83%
  Arms: Ecabet 2.83%
Drug: Ecabet 3.70%
  Arms: Ecabet 3.70%
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine whether ecabet ophthalmic solution is an effective treatment for dry eye syndrome

ELIGIBILITY:
Inclusion Criteria:

* Agree to avoid systemic & topical ophthalmic meds & disallowed meds
* Have a best corrected visual acuity (BCVA) of 20/40 with pinhole or better in each eye
* Diagnosis of moderate dry eye syndrome

Exclusion Criteria:

* Uncontrolled ocular or systemic disease that could interfere with study
* Diagnosis of Sjogren's syndrome, lacrimal obstruction, reflex, lid-related or contact lens-related dry eye syndrome(DES); significant anterior blepharitis or meibomianitis
* Contraindications or hypersensitivity to use of study meds or components
* Wear contact lenses
* Secondary dry eye to surgery
* Eye surgery (including laser) within 6 months
* Use of systemic or topical ophthalmic meds within 14 days
* Punctal plugs in one or both eyes in place for <45 days
* Permanent occlusion of the lacrimal puncta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2005-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Ocular discomfort | Day 91
  Group mean change in ocular discomfort score from pre-Cataract extraction (CAE) to post-CAE
Tear Film Break-up Time (TFBUT) | Day 91
  Group mean change in time to tear break-up from pre-CAE to post-CAE.
Blink Rate | Day 91
  Group mean change in blinks/min from pre-CAE to post-CAE.

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts
  - Eyesight Ophthalmic Services, PA, Dover, New Hampshire